CLINICAL TRIAL: NCT06984172
Title: Effectiveness of Cardiac Rehabilitation With Remote Connection Device for Patients After Surgery for Acquired Heart Valve Disease
Brief Title: Effectiveness of Remote Cardiac Rehab After Surgery for Acquired Heart Valve Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HMUIBR1880
Record Dates: First submitted 2025-05-11; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-04

CONDITIONS: Valvular Diseases
Keywords: phẫu thuật tim; phục hồi chức năng; valvular disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Undergoes acute-phase rehabilitation training for approximately 1 week immediately after surgery, then transitions to early recovery-phase rehabilitation for about another week at the hospital.
  After discharge, patients continue to be monitored and guided in their rehabilitation exercises according to the Japanese Circulation Society's protocol (2021) for 1 month (in late recovery phase) through the Open TeleRehab software.
  Physical capacity assessments are conducted at several time points: before surgery, at the end of the acute-phase rehabilitation (beginning of the early recovery phase), at hospital discharge (end of the early recovery phase), and one month after discharge.
  Interventions: Procedure: Remote cardiac rehabilitation
- Control group (Active Comparator): Undergoes acute-phase rehabilitation training for approximately 1 week immediately after surgery, then transitions to early recovery-phase rehabilitation for about another week at the hospital.
  After discharge, patients continue late-phase cardiovascular rehabilitation as outpatients for the following month.
  Physical capacity assessments are conducted at several time points: before surgery, at the end of the acute-phase rehabilitation (beginning of the early recovery phase), at hospital discharge (end of the early recovery phase), and one month after discharge.
  Interventions: Procedure: Facility-based cardiac rehabilitation

INTERVENTIONS:
Procedure: Remote cardiac rehabilitation — The patient, following heart valve surgery, is undergoing home-based cardiovascular rehabilitation during the late recovery phase. The rehabilitation is remotely supervised by a therapist through the Open TeleRehab software and includes aerobic exercises, breathing exercises, and lower limb resistance training.
  * Aerobic exercise: Performed 3 times per week, each session lasting 20-40 minutes. Activities include walking, stair climbing, or cycling. Exercise intensity is determined based on:
    1. Target heart rate: Set at the anaerobic threshold identified through Cardiopulmonary Exercise Testing (CPET) prior to hospital discharge; heart rate is monitored using a handheld pulse oximeter.
    2. Borg Rating of Perceived Exertion (RPE) scale for dyspnea: maintained at 12-13 out of 20.
  * Lower limb resistance training: Performed 3 times per week, each session lasting 30-40 minutes. Intensity is based on the one-repetition maximum (1RM).
  * Breathing exercises: Performed 3 times per week
  Other Names: home-based cardiac rehabilitation in late recovery phase
  Arms: Intervention group
Procedure: Facility-based cardiac rehabilitation — After completing inpatient rehabilitation, patients are discharged and continue supervised outpatient rehabilitation three times per week. The program includes aerobic exercise, lower limb resistance training, and breathing exercises.
  Aerobic exercise: Each session lasts 20-40 minutes, depending on the patient's condition, and is performed using a Cardiopulmonary Exercise Testing (CPET) device. Exercise intensity is determined based on the target heart rate and the Borg Rating of Perceived Exertion (RPE) scale for dyspnea and fatigue, in accordance with the 2021 guidelines of the Japanese Circulation Society.
  Lower limb resistance training: Each session lasts 30-40 minutes.
  Breathing exercises: Each session lasts 15-20 minutes
  Other Names: Late-recovery phase outpatient rehabilitation conducted at a rehabilitation center
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn if home-based cardiac rehabilitation using remote monitoring devices improves exercise capacity in patients after surgery for acquired heart valve diseases. It also aims to learn about factors affecting the outcomes of remote treatment.

The main questions it seeks to answer are:

* How does cardiac rehabilitation using remote monitoring devices improve exercise capacity in participants compared to those undergoing rehabilitation at medical facilities?
* What factors influence the outcomes of participants undergoing cardiac rehabilitation with remote monitoring devices? The researchers compare the exercise capacity of the intervention group - receiving home-based cardiac rehabilitation using remote monitoring devices - with that of the control group receiving treatment at a rehabilitation facility during the recovery phase.

All patients participating in the study receive inpatient cardiac rehabilitation during the acute phase (1 week) and the early recovery phase (1 week) at the hospital.

The control group continues supervised outpatient rehabilitation at the hospital, three sessions per week for the following month.

The intervention group undergoes home-based rehabilitation under the guidance of a therapist via the Open TeleRehab platform and self-monitors hemodynamic parameters using a personal blood pressure monitor and a handheld pulse oximeter.

Both groups are assessed for exercise capacity at baseline (pre-surgery), after each phase of rehabilitation, and one month after hospital discharge.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, single-blind interventional study. We conduct the study on patients aged 18 years and older diagnosed with acquired heart valve diseases who have an indication for valve repair or replacement surgery at the Cardiovascular Center - Hanoi Medical University Hospital.

All patients participating in the study receive inpatient cardiac rehabilitation during the acute phase (1 week) and early recovery phase (1 week) at the hospital.

Before discharge, patients are randomly assigned by dice rolling into the intervention or control group, with a minimum of 22 patients in each group.

The control group continues supervised outpatient rehabilitation at the hospital, three sessions per week for the following month.

The intervention group undergoes home-based rehabilitation and self-monitors their hemodynamic parameters using a personal blood pressure monitor and a handheld pulse oximeter. Before and after each training session, patients send images of their vital signs (heart rate, blood pressure, SpO₂) to the physician via the Open TeleRehab platform. The physician immediately provides feedback if adjustments to the exercise session (intensity, duration, type) are necessary.

Every Saturday, physicians and patients conduct a group meeting via the Open TeleRehab platform to discuss any issues arising during the training sessions (approximately 30 minutes).

Exercise capacity assessments for both groups are performed at baseline (pre-surgery), after acute phase rehabilitation, before discharge, and one month post-discharge.

Evaluation parameters include: 6-minute walk distance, 2-minute step test, and peak oxygen uptake (VO₂ peak) measured by cardiopulmonary exercise testing (CPET).

Cardiac rehabilitation interventions are conducted following the 2021 guidelines of the Japanese Circulation Society.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing first-time surgery for acquired heart valve diseases (valve replacement or repair), including the aortic valve, mitral valve, tricuspid valve, pulmonary valve, or a combination of these valves.
* Willing to participate in the study.

Exclusion Criteria:

* Contraindications to cardiac rehabilitation.
* Patients who die during the study after hospital discharge.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen uptake | At the beginning of the early recovery phase (typically around 10 days after surgery), at the end of the early rehabilitation phase (immediately before hospital discharge), and one month later
  Maximal oxygen uptake (VO₂ max) refers to the maximum amount of oxygen that an individual can utilize during intense or maximal exercise. And it is a gold standard indicator of cardiovascular and respiratory system efficiency.
  VO₂ max is typically measured using cardiopulmonary exercise testing (CPET). Higher VO₂ max values are associated with better cardiovascular health, lower risk of heart disease, and greater endurance.
Six-Minute Walk Test | pre-operation, at the beginning of the early recovery phase, at the end of the early rehabilitation phase, and one month later
  Six-Minute Walk Test (6MWT) is used widely due to its simplicity and reproducibility, delivering a consolidated image of the cardiopulmonary and musculoskeletal response to exercise.
  This test accurately measures the maximum distance a person can walk in 6 minutes. It requires only simple, commonly available equipment such as a pulse oximeter, a portable oxygen device (to be used if needed by the patient), a chair, a validated dyspnea scale (e.g., the Borg scale), and a stopwatch.
  However, the study cannot identify the cause of dyspnea, or hypoxemia, or the mechanisms underlying a particular patient's exercise intolerance. Because of this, we conduct both 6MWT and Cardiopulmonary Exercise Testing (CPET) on this research.
  Among healthy individuals, the average 6MWT is between 400 and 700 meters.

SECONDARY OUTCOMES:
Two-minute Step Test | pre-operation, at the beginning of the early recovery phase, at the end of the early rehabilitation phase, and one month later
  The 2-minute step test is one of the physical capacity assessments, introduced since 1999. The advantages of TMST are that it is safe, does not require a large space, is quick to perform and does not require expensive equipment, has high test-retest reliability (0.9 - Rikli's study), is highly sensitive, and has a small learning effect. Disadvantages: the implementation method is inconsistent in previous studies (some studies count the number of steps of both legs, some studies only count the number of steps of the right leg).
  TMST has been studied and shown to correlate well with other physical capacity assessments such as 1-mile walking time, 6MWT. The results differ between age groups and genders How to perform (as first described by Rikli): count the number of times the patient steps in place, raising the knee to the midpoint of the line connecting the iliac crest to the patella, in 2 minutes. In this study, the assessor counted the number of steps that met the standard for both

CONTACTS AND LOCATIONS:
Overall Officials: Phạm Văn Minh, Assoc. Prof. MD, Principal Investigator — Trường Đại học Y Hà Nội; Vũ Ngọc Tú, Assoc. Prof. MD, Principal Investigator — Trường Đại học Y Hà Nội
Locations (1):
- Hanoi Medical University Hospital, Hà Nội, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bohannon RW, Crouch RH. Two-Minute Step Test of Exercise Capacity: Systematic Review of Procedures, Performance, and Clinimetric Properties. J Geriatr Phys Ther. 2019 Apr/Jun;42(2):105-112. doi: 10.1519/JPT.0000000000000164. PMID 29210933
- [Background] Agarwala P, Salzman SH. Six-Minute Walk Test: Clinical Role, Technique, Coding, and Reimbursement. Chest. 2020 Mar;157(3):603-611. doi: 10.1016/j.chest.2019.10.014. Epub 2019 Nov 2. PMID 31689414
- [Background] Pritchard A, Burns P, Correia J, Jamieson P, Moxon P, Purvis J, Thomas M, Tighe H, Sylvester KP. ARTP statement on cardiopulmonary exercise testing 2021. BMJ Open Respir Res. 2021 Nov;8(1):e001121. doi: 10.1136/bmjresp-2021-001121. PMID 34782330
- [Background] Razvi Y, Ladie DE. Cardiopulmonary Exercise Testing. 2023 Apr 24. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK557886/ PMID 32491809
- [Background] Adachi H. Cardiopulmonary Exercise Test. Int Heart J. 2017 Oct 21;58(5):654-665. doi: 10.1536/ihj.17-264. Epub 2017 Sep 30. PMID 28966333
- [Background] McDonagh ST, Dalal H, Moore S, Clark CE, Dean SG, Jolly K, Cowie A, Afzal J, Taylor RS. Home-based versus centre-based cardiac rehabilitation. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD007130. doi: 10.1002/14651858.CD007130.pub5. PMID 37888805
- [Background] Hansen TB, Zwisler AD, Berg SK, Sibilitz KL, Thygesen LC, Kjellberg J, Doherty P, Oldridge N, Sogaard R. Cost-utility analysis of cardiac rehabilitation after conventional heart valve surgery versus usual care. Eur J Prev Cardiol. 2017 May;24(7):698-707. doi: 10.1177/2047487317689908. Epub 2017 Jan 25. PMID 28121172
- [Background] Li Z, Song W, Yang N, Ding Y. Exercise-based cardiac rehabilitation programmers for patients after transcatheter aortic valve implantation: A systematic review and meta-analysis. Medicine (Baltimore). 2023 Jul 28;102(30):e34478. doi: 10.1097/MD.0000000000034478. PMID 37505146
- [Background] Pavy B, Iliou MC, Meurin P, Tabet JY, Corone S; Functional Evaluation and Cardiac Rehabilitation Working Group of the French Society of Cardiology. Safety of exercise training for cardiac patients: results of the French registry of complications during cardiac rehabilitation. Arch Intern Med. 2006 Nov 27;166(21):2329-34. doi: 10.1001/archinte.166.21.2329. PMID 17130385
- [Background] Tessler J, Ahmed I, Bordoni B. Cardiac Rehabilitation. 2025 Mar 28. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK537196/ PMID 30725881
- [Background] Kang YR, Kim JS, Cha YK, Jeong YJ. Imaging findings of complications after thoracic surgery. Jpn J Radiol. 2019 Mar;37(3):209-219. doi: 10.1007/s11604-018-00806-y. Epub 2019 Jan 12. PMID 30637569
- [Background] Popovici M, Ursoniu S, Feier H, Mocan M, Tomulescu OMG, Kundnani NR, Valcovici M, Dragan SR. Benefits of Using Smartphones and Other Digital Methods in Achieving Better Cardiac Rehabilitation Goals: A Systematic Review and Meta-Analysis. Med Sci Monit. 2023 May 5;29:e939132. doi: 10.12659/MSM.939132. PMID 37143317
- [Background] Aluru JS, Barsouk A, Saginala K, Rawla P, Barsouk A. Valvular Heart Disease Epidemiology. Med Sci (Basel). 2022 Jun 15;10(2):32. doi: 10.3390/medsci10020032. PMID 35736352
- [Result] Dorje T, Zhao G, Tso K, Wang J, Chen Y, Tsokey L, Tan BK, Scheer A, Jacques A, Li Z, Wang R, Chow CK, Ge J, Maiorana A. Smartphone and social media-based cardiac rehabilitation and secondary prevention in China (SMART-CR/SP): a parallel-group, single-blind, randomised controlled trial. Lancet Digit Health. 2019 Nov;1(7):e363-e374. doi: 10.1016/S2589-7500(19)30151-7. Epub 2019 Oct 10. PMID 33323210
- [Result] Lunde P, Bye A, Bergland A, Grimsmo J, Jarstad E, Nilsson BB. Long-term follow-up with a smartphone application improves exercise capacity post cardiac rehabilitation: A randomized controlled trial. Eur J Prev Cardiol. 2020 Nov;27(16):1782-1792. doi: 10.1177/2047487320905717. Epub 2020 Feb 28. PMID 32106713
- [Result] Sibilitz KL, Tang LH, Berg SK, Thygesen LC, Risom SS, Rasmussen TB, Schmid JP, Borregaard B, Hassager C, Kober L, Taylor RS, Zwisler AD. Long-term effects of cardiac rehabilitation after heart valve surgery - results from the randomised CopenHeartVR trial. Scand Cardiovasc J. 2022 Dec;56(1):247-255. doi: 10.1080/14017431.2022.2095432. PMID 35811477
- [Result] Makita S, Yasu T, Akashi YJ, Adachi H, Izawa H, Ishihara S, Iso Y, Ohuchi H, Omiya K, Ohya Y, Okita K, Kimura Y, Koike A, Kohzuki M, Koba S, Sata M, Shimada K, Shimokawa T, Shiraishi H, Sumitomo N, Takahashi T, Takura T, Tsutsui H, Nagayama M, Hasegawa E, Fukumoto Y, Furukawa Y, Miura SI, Yasuda S, Yamada S, Yamada Y, Yumino D, Yoshida T, Adachi T, Ikegame T, Izawa KP, Ishida T, Ozasa N, Osada N, Obata H, Kakutani N, Kasahara Y, Kato M, Kamiya K, Kinugawa S, Kono Y, Kobayashi Y, Koyama T, Sase K, Sato S, Shibata T, Suzuki N, Tamaki D, Yamaoka-Tojo M, Nakanishi M, Nakane E, Nishizaki M, Higo T, Fujimi K, Honda T, Matsumoto Y, Matsumoto N, Miyawaki I, Murata M, Yagi S, Yanase M, Yamada M, Yokoyama M, Watanabe N, Itoh H, Kimura T, Kyo S, Goto Y, Nohara R, Hirata KI; Japanese Circulation Society/the Japanese Association of Cardiac Rehabilitation Joint Working Group. JCS/JACR 2021 Guideline on Rehabilitation in Patients With Cardiovascular Disease. Circ J. 2022 Dec 23;87(1):155-235. doi: 10.1253/circj.CJ-22-0234. Epub 2022 Dec 9. No abstract available. PMID 36503954
- [Result] Xue W, Xinlan Z, Xiaoyan Z. Effectiveness of early cardiac rehabilitation in patients with heart valve surgery: a randomized, controlled trial. J Int Med Res. 2022 Jul;50(7):3000605211044320. doi: 10.1177/03000605211044320. PMID 35899970

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT06984172/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT06984172/ICF_001.pdf